CLINICAL TRIAL: NCT05021250
Title: Stereotactic Body Radiation Therapy With Deep Inspiration Breath Hold for Hepatocellular Carcinoma After Transcatheter Arterial Chemoembolization and Lipiodol Marking
Brief Title: SBRT With DIBH for HCC After TACE and Lipiodol Marking
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: The First Hospital of Jilin University (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, BO CHEN, Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC2713
Record Dates: First submitted 2021-06-23; First posted 2021-08-25 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma, TACE, SBRT, DIBH
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: HCC patients treated with TACE and lipiodol marking, followed by SBRT with DIBH which was registrated with lipiodol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lipiodol marking (Experimental): HCC patients treated with TACE and lipiodol marking, followed by SBRT with DIBH.
  Interventions: Procedure: Lipiodol marking

INTERVENTIONS:
Procedure: Lipiodol marking — HCC patients treated with TACE and the tumor marked with lipiodol.

SUMMARY:
Stereotactic Body Radiation Therapy (SBRT) for hepatocellular carcinoma (HCC) with radical dose achieved similar results with radiofrequency ablation (RF) and radical surgery, according to previous studies. For tumors near great blood vessels or with a diameter more than 2cm, SBRT performs even better than RF. In current clinical practice of SBRT for small HCC, registration is achieved by planting metal markers near the tumor, which has several disadvantages: 1. the operation is invasive, increase the risk of bleeding in patients with cirrhosis; 2. the operation is of no therapeutic value; 3. metal markers can only be planted outside the tumor to avoid transplantation, which compromises the accuracy of registration via CBCT. This study aims to adopt a new method of registration, transcatheter arterial chemoembolization (TACE) and lipiodol marking, to analyze the recognition and clarity of lipiodol on CBCT images, set-up errors and treatment efficacy. Therefore to provide data to support TACE and lipiodol marking over metal marker planting.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically or pathologically confirmed hepatocellular carcinoma.
2. ECOG 0-1.
3. BCLC C
4. Liver-GTV >700ml; intrahepatic metastasis allowed but only one tumor is to be treated with SBRT and others stable for more than 3 months; distant metastasis allowed but stable for more than 6 months.
5. Expected gastric/duodenum/small intestine Dmax 25-35Gy; colon Dmax 28-38Gy. Prescription dose 40Gy/5-10f.
6. DIBH training prior to SBRT to achieve 36 seconds breath hold.
7. Life expectancy > 3 months.
8. Child-Pugh A5, A6 or B7.
9. Liver function: ALT within 1.5 times of upper limit; ALT within 0.5 times of upper limit and AST within 6 times of upper limit, excluding cardiac infarction; ALT within 0.5-1.5 times of upper limit and AST within 1.5 times of upper limit
10. Normal ECG, without severe cardiac dysfunction
11. Kidney function: CRE, BUN within 1.5 times of upper limit.
12. CBC: Hb≥80g/L，ANC≥1.0×109 /L，PLT≥40×109 /L
13. Without hemorrhagic tendency.
14. Voluntarily participate in this trial and sign consent form.

Exclusion Criteria:

1. Participants of other clinical trials.
2. History of abdomen radiation therapy or liver transplantation.
3. History of severe cardiovascular, kidney or liver disease.
4. Pregnancy or lactation.
5. Suspected or confirmed of drug or alcohol abuse.
6. History of severe mental or neurological disease, compromising the ability to consent and/or AE diagnosis.
7. Allergic to lipiodol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Recognition of lipiodol marking | During the radiotherapy
  Judged by 2 technicians and 1 physician on CBCT images. High recognition is concluded when all three consider it easily registered. Moderate recognition is concluded when two consider it easily registered. Poor recognition is concluded when one or none consider it easily registered.
ORR | 6 months after radiotherapy
  Objective response rate

SECONDARY OUTCOMES:
Completion rate of treatment model | 1 months after TACE
  Including the success rate of lipiodol deposition at 1 months after TACE and completion of SBRT
LCR | 12 months and 24 months after radiotherapy
  Local control rate
PFS | 12 months and 24 months after radiotherapy
  Progress free survival
Frequency of AE | up to 24 months
  Frequency of treatment associated adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bo Chen, Principal Investigator — National Cancer Center/Cancer Hospital
Locations (1):
- Bo Chen, Beijing, Beijing Municipality, China